CLINICAL TRIAL: NCT00620399
Title: Lumbar Fusion With and Without Postoperative Bracing: A Randomized Prospective Study
Brief Title: A Study on the Use of a Brace Following Low Back Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Medtronic Sofamor Danek (Unknown)
Responsible Party: Sanford Emery and Albert Yee, Sunnybrook Health Sciences Centre
Purpose: Treatment
Other Study IDs: 019511
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Lumbar Fusion
Keywords: lumbar fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): brace
  Interventions: Other: lumbar corset
- 2 (Placebo Comparator): no brace
  Interventions: Other: lumbar corset

INTERVENTIONS:
Other: lumbar corset

SUMMARY:
This study evaluated the hypothesis that bracing following lumbar spinal fusion surgery improves functional outcome following surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Undergoing posterior lumbar fusion surgery for degenerative conditions

Exclusion Criteria:

* Unable to complete questionnaires due to language or cognitive barrier
* Declined study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-05; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
functional outcome scores | 2 years following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States